CLINICAL TRIAL: NCT04560062
Title: Contextualizing Evidence for Action on Diabetes in Low-resource Settings: a Mixed-methods Case Study in Quito and Esmeraldas, Ecuador.
Brief Title: Contextualizing the Evidence for Action on Diabetes - Cohort
Acronym: CEAD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universidad Miguel Hernandez de Elche (Other)
Collaborators: European Research Council (Other); Pontificia Universidad Católica del Ecuador (Unknown); Centro de Epidemiología Comunitaria y Medicina Tropical (Unknown)
Responsible Party: Principal Investigator, Lucy Anne Parker, Lecturer, Universidad Miguel Hernandez de Elche
Other Study IDs: ERC-2018-STG-804761.2
Record Dates: First submitted 2020-08-27; First posted 2020-09-23 (Actual); Last update posted 2021-01-25 (Actual); Status verified 2021-01

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Implementation science; Delivery of Health Care; Public Policy; Non-communicable Disease
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Noncommunicable Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Population in Quito: 576 randomly chosen patients with diabetes in District 17D06, Quito (Ecuador)
  Interventions: Other: Spontaneous changes in diabetes-related health care
- Population in Esmeraldas: 576 randomly chosen patients with diabetes in Eloy Alfaro District, Esmeraldas (Ecuador)
  Interventions: Other: Spontaneous changes in diabetes-related health care

INTERVENTIONS:
Other: Spontaneous changes in diabetes-related health care — The findings of a retrospective cohort analysis conducted in the initial phase of the study will be used in focus groups to identify observed weaknesses in local health systems and will promote possible solutions to strengthen diabetes-related health care. Every focus group will include community members, healthcare workers, decision-makers and diabetic patients and family members.

SUMMARY:
This protocol reflects the second part of a larger mixed-methods study aimed at exploring the process by which global recommendations can be translated into context-specific, evidence-informed action for diabetes prevention in low-resource settings. Firstly, a retrospective cohort study will assess the current level of implementation of comprehensive diabetes care over a 24-month period (2019-2020), by describing healthcare received and health outcomes of a representative sample of diabetes patients currently accessing care in the study region. Focus groups prompted by the findings of the retrospective study will be used to inspire local innovations which will be evaluated through a prospective follow-up of the cohort.

DETAILED DESCRIPTION:
Objective: To evaluate the implementation of comprehensive diabetes care in two low-resource settings in Ecuador.

Specific objectives:

1. To assess patient outcomes including biochemical diabetes control and health-related quality of life.
2. To evaluate diabetes-related health care access.
3. To assess complications related to diabetes.

Sample size: The sample size is proposed conservatively to ensure a precision to estimate outcomes of 50% with an absolute precision of ±5%, assuming a design effect of 1.2 and potential loss of 20%.

Sample design: A representative sample for each district will be obtained by stratified single-stage cluster sampling. The clusters are health facilities for which a sample of patients will randomly selected. The sample will be stratified by facility type (Ministry of Public Health (MSP) facilities, or Social Security facilities for affiliated workers) in Quito and by Rural/Urban setting in Esmeraldas. Patient sampling will use the electronic consultation registry of each selected facility where possible. Data unavailable in the electronic registers will be extracted from any available paper files.

Data collection procedure: Research assistants will obtain the data mainly from health services records, which will be supplemented by patient interviews including socio-demographic and clinical data, perceived social support (the Multidimensional Scale of Perceived Social Support, MSPSS) and health-related quality of life (the Diabetes Health Profile-18, DHP-18) profile. They will collect data regarding whether the patient received regular review by a clinician, and underwent screening for diabetes complications as recommended in the 2017 Clinical Practice Guideline for Type 2 Diabetes in Ecuador. He/she will record the date and details of any complications and experiences over the course of the evaluation and other clinical data such as comorbidities, treatments or patient management by a multidisciplinary health care team.

The first data collection will be retrospective and will include diabetes-related health care and clinical outcomes during 2019 and 2020. Clinical files will be reviewed every 12 months for the duration of follow-up (2 years). Supplementary interview data will be assessed on a baseline and in the last 6 months of follow-up.

Analysis: The researchers will calculate the proportion of patients that received care as per the clinical practice guideline (CPG) recommendations and/or the proportion receiving an intermediate level of care (as required). Proportions will be described with 95% confidence intervals. Variation in healthcare received and diabetes-related health will be described using sociodemographic and clinical characteristics of the patients to highlight potential inequities. A multivariate logistic regression model may be used to explore the relationship between the primary outcomes and socioeconomic explanatory variable and/or type of health facility. If necessary, the researchers will adjust for potential confounders such as patients' factors (e.g. sex, age, comorbidity, perceived social support) and/or environmental factors (e.g. proximity to the health centre, availability of different medical specialties or methods as laboratory test). Statistical analysis will be performed using Stata/SE (StataCorp, College Station, TX, USA) Version 15.

ELIGIBILITY:
Inclusion Criteria:

* Individuals diagnosed with type-2 diabetes.
* Age over 18 years.
* Patients are accessing diabetes care in health facilities in the study districts.
* Providing informed consent

Exclusion Criteria:

* Unability to provide informed consent (e.g. significant mental impairment).
* Pregnant women if they are diagnosed with gestational diabetes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The CEAD project will be carried out in 2 low-resource settings in Ecuador: 1) District 17D06, South Quito, an urban health district ; and 2) District 08D02, Eloy Alfaro District, in Esmeraldas Province, a rural area in the northern coastal region of the country.
Sampling Method: Probability Sample
Enrollment: 1152 (Estimated)
Dates: Start 2020-10-13 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with biochemically controlled disease | Year 1
  Proportions of patients with controlled disease along with 95% confidence interval.
  Controlled disease is defined according to the last laboratory result as glycated haemoglobin <7% or <8% if ≥15 years of evolution or complications and serious comorbidities; or fasting blood glucose: 70 - 130 mg/dl or postprandial blood glucose <180 mg/dl.
Proportion of patients with biochemically controlled disease | Year 2
  Proportions of patients with controlled disease along with 95% confidence interval.
  Controlled disease is defined according to the last laboratory result as glycated haemoglobin <7% or <8% if ≥15 years of evolution or complications and serious comorbidities; or fasting blood glucose: 70 - 130 mg/dl or postprandial blood glucose <180 mg/dl.
Proportion of patients with biochemically controlled disease | Year 3
  Proportions of patients with controlled disease along with 95% confidence interval.
  Controlled disease is defined according to the last laboratory result as glycated haemoglobin <7% or <8% if ≥15 years of evolution or complications and serious comorbidities; or fasting blood glucose: 70 - 130 mg/dl or postprandial blood glucose <180 mg/dl.
Proportion of patients with biochemically controlled disease | Year 4
  Proportions of patients with controlled disease along with 95% confidence interval.
  Controlled disease is defined according to the last laboratory result as glycated haemoglobin <7% or <8% if ≥15 years of evolution or complications and serious comorbidities; or fasting blood glucose: 70 - 130 mg/dl or postprandial blood glucose <180 mg/dl.
Proportion of patients with optimal health-related quality of life | Year 3
  Health-related quality of life will be obtained with Diabetes Health Profile-18 (DHP-18) questionnaire. DHP-18 scores range from 0 to 100, with 0 representing no dysfunction and 100 maximum dysfunction.
  Proportion of patients with total final score under the median, meaning lower dysfunction, along with 95% confidence interval.
Proportion of patients with optimal health-related quality of life | Year 4
  Health-related quality of life will be obtained with Diabetes Health Profile-18 (DHP-18) questionnaire. DHP-18 scores range from 0 to 100, with 0 representing no dysfunction and 100 maximum dysfunction.
  Proportion of patients with total final score under the median, meaning lower dysfunction, along with 95% confidence interval.
Proportion of patients with access to health care of diabetes | Year 1
  It includes processes of care indicators that represent the proportion of the patients who undergo the care processes recommended by the CPG to manage the disease. The investigators will obtain the care frequency for each patient during the year of study as a quantitative value and will also categorize those care indicators that are recommended with greater periodicity in the CPG.
Proportion of patients with access to health care of diabetes | Year 2
  It includes processes of care indicators that represent the proportion of the patients who undergo the care processes recommended by the CPG to manage the disease. The investigators will obtain the care frequency for each patient during the year of study as a quantitative value and will also categorize those care indicators that are recommended with greater periodicity in the CPG.
Proportion of patients with access to health care of diabetes | Year 3
  It includes processes of care indicators that represent the proportion of the patients who undergo the care processes recommended by the CPG to manage the disease. The investigators will obtain the care frequency for each patient during the year of study as a quantitative value and will also categorize those care indicators that are recommended with greater periodicity in the CPG.
Proportion of patients with access to health care of diabetes | Year 4
  It includes processes of care indicators that represent the proportion of the patients who undergo the care processes recommended by the CPG to manage the disease. The investigators will obtain the care frequency for each patient during the year of study as a quantitative value and will also categorize those care indicators that are recommended with greater periodicity in the CPG.

SECONDARY OUTCOMES:
Perceived social support | Year 3
  Results of the standardized questionnaire "the Multidimensional Scale of Perceived Social Support (MSPSS)". The response format is a four-point Likert type scale (1= rarely, 2= sometimes, 3=frequently, 4= always or almost always). A higher score implies a greater perception of social support.
  Tertiles of total final score will be used to measure low, medium and high social support. The investigators will report the patient ratio and 95% confidence interval for each category of social support
Perceived social support | Year 4
  Results of the standardized questionnaire "the Multidimensional Scale of Perceived Social Support (MSPSS)". The response format is a four-point Likert type scale (1= rarely, 2= sometimes, 3=frequently, 4= always or almost always). A higher score implies a greater perception of social support.
  Tertiles of total final score will be used to measure low, medium and high social support. The investigators will report the patient ratio and 95% confidence interval for each category of social support.
Proportion of patients who diabetes-related education received | Year 3
  Self-reported information [dichotomous (yes/no) responses]. Proportion of patients who indicate that they have received information on diabetes and healthy habits, along with 95% confidence interval.
Proportion of patients who diabetes-related education received | Year 4
  Self-reported information [dichotomous (yes/no) responses]. Proportion of patients who indicate that they have received information on diabetes and healthy habits, along with 95% confidence interval.
Proportion of patients with blood pressure controlled (<140/90 mmHg) | Year 1
  Proportions along with 95% confidence interval.
Proportion of patients with blood pressure controlled (<140/90 mmHg) | Year 2
  Proportions along with 95% confidence interval.
Proportion of patients with blood pressure controlled (<140/90 mmHg) | Year 3
  Proportions along with 95% confidence interval.
Proportion of patients with blood pressure controlled (<140/90 mmHg) | Year 4
  Proportions along with 95% confidence interval.
Proportion of patients with BMI between 18.5 and 25 kg/m2 or 5% weight loss if BMI>25 kg/m2 | Year 1
  Proportions along with 95% confidence interval.
Proportion of patients with BMI between 18.5 and 25 kg/m2 or 5% weight loss if BMI>25 kg/m2 | Year 2
  Proportions along with 95% confidence interval.
Proportion of patients with BMI between 18.5 and 25 kg/m2 or 5% weight loss if BMI>25 kg/m2 | Year 3
  Proportions along with 95% confidence interval.
Proportion of patients with BMI between 18.5 and 25 kg/m2 or 5% weight loss if BMI>25 kg/m2 | Year 4
  Proportions along with 95% confidence interval.
Proportion of patients with LDL cholesterol level < 100 mg/dl | Year 1
  Proportions along with 95% confidence interval.
Proportion of patients with LDL cholesterol level < 100 mg/dl | Year 2
  Proportions along with 95% confidence interval.
Proportion of patients with LDL cholesterol level < 100 mg/dl | Year 3
  Proportions along with 95% confidence interval.
Proportion of patients with LDL cholesterol level < 100 mg/dl | Year 4
  Proportions along with 95% confidence interval.
Proportion of patients with microalbuminuria level <30 mg/day | Year 1
  Proportions along with 95% confidence interval.
Proportion of patients with microalbuminuria level <30 mg/day | Year 2
  Proportions along with 95% confidence interval.
Proportion of patients with microalbuminuria level <30 mg/day | Year 3
  Proportions along with 95% confidence interval.
Proportion of patients with microalbuminuria level <30 mg/day | Year 4
  Proportions along with 95% confidence interval.
Number of unscheduled diabetes-related consultations | Year 1
  Number of unscheduled due to decompensation of the disease and/or complications. Results will be reported as absolute values.
Number of unscheduled diabetes-related consultations | Year 2
  Number of unscheduled due to decompensation of the disease and/or complications. Results will be reported as absolute values.
Number of unscheduled diabetes-related consultations | Year 3
  Number of unscheduled due to decompensation of the disease and/or complications. Results will be reported as absolute values.
Number of unscheduled diabetes-related consultations | Year 4
  Number of unscheduled due to decompensation of the disease and/or complications. Results will be reported as absolute values.
Number of hospitalisations due to diabetes complications | Year 1
  Number of hospitalisations owing to decompensation of the disease and/or complications. Results will be reported as absolute values.
Number of hospitalisations due to diabetes complications | Year 2
  Number of hospitalisations owing to decompensation of the disease and/or complications. Results will be reported as absolute values.
Number of hospitalisations due to diabetes complications | Year 3
  Number of hospitalisations owing to decompensation of the disease and/or complications. Results will be reported as absolute values.
Number of hospitalisations due to diabetes complications | Year 4
  Number of hospitalisations owing to decompensation of the disease and/or complications. Results will be reported as absolute values.
Proportion of patients with at least one disease complication | Year 1
  Disease complications considered will include retinopathy and/or blindness, lower limb amputations, cardiovascular events (such as stroke, myocardial infarction, ischemic heart disease, obstructive artery disease, congestive heart failure) and/or renal dysfunction according to the last glomerular filtration rate result using the MDRD-4 (Modification of Diet in Renal Disease) formula or serum creatinine value.
  Proportion along with 95% confidence interval.
Proportion of patients with at least one disease complication | Year 2
  Disease complications considered will include retinopathy and/or blindness, lower limb amputations, cardiovascular events (such as stroke, myocardial infarction, ischemic heart disease, obstructive artery disease, congestive heart failure) and/or renal dysfunction according to the last glomerular filtration rate result using the MDRD-4 (Modification of Diet in Renal Disease) formula or serum creatinine value.
  Proportion along with 95% confidence interval.
Proportion of patients with at least one disease complication | Year 3
  Disease complications considered will include retinopathy and/or blindness, lower limb amputations, cardiovascular events (such as stroke, myocardial infarction, ischemic heart disease, obstructive artery disease, congestive heart failure) and/or renal dysfunction according to the last glomerular filtration rate result using the MDRD-4 (Modification of Diet in Renal Disease) formula or serum creatinine value.
  Proportion along with 95% confidence interval.
Proportion of patients with at least one disease complication | Year 4
  Disease complications considered will include retinopathy and/or blindness, lower limb amputations, cardiovascular events (such as stroke, myocardial infarction, ischemic heart disease, obstructive artery disease, congestive heart failure) and/or renal dysfunction according to the last glomerular filtration rate result using the MDRD-4 (Modification of Diet in Renal Disease) formula or serum creatinine value.
  Proportion along with 95% confidence interval.

CONTACTS AND LOCATIONS:
Overall Officials: Lucy A Parker, PhD, Principal Investigator — University Miguel Hernández
Locations (1):
- Mari Carmen Bernal Soriano, Esmeraldas, Ecuador

IPD SHARING:
Plan to Share IPD: Yes
This research is part of a European Research Council Grant and we are participating in the Open Data Research Plan.
Supporting Information: Study Protocol, SAP
Time Frame: The study protocol will by published in an open access journal within the first 6 months of study recruitment. The Statistical Analysis Plan will be available before study recruitment is completed.
Access Criteria: Open Access